CLINICAL TRIAL: NCT06965894
Title: Effect of Pressure Splints on Lower Extremity Functions in Hemiplegic Stroke Patients
Brief Title: Lower Extremity Pressure Splints in HP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Çiçek Günday, Asst. Prof., Istinye University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 02052025
Record Dates: First submitted 2025-04-30; First posted 2025-05-11 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Hemiplegia; Lower Extremity Dysfunction; Stroke Rehabilitation
Keywords: Stroke; Rehabilitation; Gait; Johnstone Splint; Motor Recovery
MeSH Terms: conditions — Hemiplegia; Stroke | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splint Group (Experimental): Participants in this group will receive a rehabilitation program including neurodevelopmental therapy and proprioceptive neuromuscular facilitation (PNF) techniques. In addition to the rehabilitation program, a Johnston pressure splint will be applied to the affected lower extremity during therapy sessions. The intervention aims to provide controlled pressure and support to improve motor recovery, balance, and gait in hemiplegic stroke patients.
  Interventions: Device: Johnston Pressure Splint; Other: Rehabilitation Program
- Control Group (Active Comparator): Participants in this group will receive a rehabilitation program including neurodevelopmental therapy and proprioceptive neuromuscular facilitation (PNF) techniques without the pressure splint. This group will serve to compare the effects of standard rehabilitation alone versus rehabilitation combined with pressure splinting.
  Interventions: Other: Rehabilitation Program

INTERVENTIONS:
Device: Johnston Pressure Splint — Application of a Johnston pressure splint to the lower extremity.
  Arms: Splint Group
Other: Rehabilitation Program — Rehabilitation program including neurodevelopmental therapy and proprioceptive neuromuscular facilitation (PNF) techniques.

SUMMARY:
Hemiplegia (weakness or paralysis on one side of the body) often impacts the lower extremities, making it challenging for patients to walk or move their legs effectively. This study aims to explore the effects of pressure splints on the lower extremity movement and function in individuals who have experienced a stroke and suffer from hemiplegia. Pressure splints are specialized devices designed to support and enhance muscle function by applying gentle pressure to the affected limbs.

Participants in this study will be randomly assigned to one of two groups: the Splint Group (SG) or the Control Group (CG). The duration of the intervention will be six weeks. During this period, all the participants will receive neurodevelopmental therapy. In the SG exercises will be done with the help of the lower extremity pressure splints while participants in the CG will join the exercises without any splint.

This study is significant as it may lead to the development of new methods to enhance recovery for stroke patients and offer better rehabilitation options.

ELIGIBILITY:
Inclusion Criteria:

* Having hemiplegia because of stroke
* Time since stroke: 1 month to 1 year
* Ability to Participate (a score of >24 on the Mini-Mental State Examination).
* Being voluntary
* Age between 50-80

Exclusion Criteria:

Severe Cognitive Impairment Other Neurological Disorders Severe Comorbidities or Spasticity on Lower Extremity Contraindications to Exercise Recurrent Stroke

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-05-13 (Actual); Primary Completion 2026-01-13 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
Lower Extremity Motor Function | Through study completion, an average of 8 months
  The improvement in motor function of the lower extremity will be assessed by Fugl-Meyer Assessment for Lower Extremity (FMA). The FMA is a stroke-specific, performance-based impairment index. It is designed to assess motor functioning, balance, sensation and joint functioning in patients with post-stroke hemiplegia. Scoring is based on direct observation of performance. Scale items are scored on the basis of ability to complete the item using a 3-point ordinal scale where 0=cannot perform, 1=performs partially and 2=performs fully. The total possible scale score is 34.
Balance | Through study completion, an average of 8 months
  The Berg Balance Scale (BBS) will be used to assess balance. This scale objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete.
Lower Extremity Strength | Through study completion, an average of 8 months
  The Five Times Sit to Stand Test will be used for the assessment of lower limb strength along with balance and postural control. Score is the amount of time it takes for an patient to transfer from a seated position to standing position and back to sitting five times.
Mobility | Through study completion, an average of 8 months
  Mobility will be assessed by Timed Up and Go (TUG). TUG is a simple test used to assess a person's mobility and requires both static and dynamic balance. It uses the time that a person takes to rise from a chair, walk three meters, turn around 180 degrees, walk back to the chair, and sit down while turning 180 degrees.

SECONDARY OUTCOMES:
Stroke Recovery | Through study completion, an average of 8 months
  The lower extremity recovery will be assessed by Brunnstrom Recovery Stages (BRS). The BRS is the most commonly used staging scale for limb function recovery in post-stroke patients. The BRS assessment scores the clinical severity of hemiplegia from 1 to 6. A score of 1 indicates paralysis and 6 indicates normal force and function
Ambulation | Through study completion, an average of 8 months
  The patients' ambulation will be assessed using the Functional Ambulation Category (FAC). FAC evaluates ambulation in 6 categories ranging from 0 to 5. A score of 0 means that the patient is not ambulatory, and 5 indicates normal ambulation.
Independence | Through study completion, an average of 8 months
  Independence will be assessed by the Functional Independence Measure (FIM). FIM is one of the most highly recommended tools for assessing functional recovery in stroke patients. This tool is considered reliable and has been proven to possess high validity for measuring the functional outcomes of stroke patients. FIM consists of 18 items related to daily activities, with a total score ranging from 18 to 126. Each item is rated on a 7-point scale, ranging from 1 (completely dependent) to 7 (independent), based on the level of independence. A total score of ≤108 indicates the need for assistance or limitations in activities.
Muscle Tone | Through study completion, an average of 8 months
  The Muscle Tone of Quadriceps and Gastrocnemius will be measured by using Modified Ashworth Scale. Modified Ashworth Scale tool used to measure the increase of muscle tone in stroke patients. The original Ashworth scale was a 5 point numerical scale that graded spasticity from 0 to 4, with 0 being no resistance and 4 being a limb rigid in flexion or extension.

CONTACTS AND LOCATIONS:
Overall Officials: Mansour Dib, Doctor, Study Chair — Mgr Cortbawi Hospital
Locations (1):
- Monseigneur Cortbawi Hospital, Jounieh, Keserwan, Lebanon

IPD SHARING:
Plan to Share IPD: No